CLINICAL TRIAL: NCT05460611
Title: A Pilot Study Evaluating the Safety and Efficacy of a 1470nm Laser for the Treatment of Androgenetic Alopecia and Scarring Alopecia
Brief Title: 1470nm Laser for the Treatment of Androgenetic Alopecia and Scarring Alopecia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14192
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Scarring Alopecia; Androgenetic Alopecia
Keywords: alopecia; laser
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Androgenetic Alopecia (Experimental): The parameters of the laser will be set according to optimal operation protocol and in accordance with guidelines set forth by Sciton. Each laser treatment will take approximately 10 to 15 minutes per subject to target androgenetic alopecia.
  Interventions: Device: Sciton HALO 1470nm Non-ablative laser
- Scarring Alopecia (Experimental): The parameters of the laser will be set according to optimal operation protocol and in accordance with guidelines set forth by Sciton. Each laser treatment will take approximately 10 to 15 minutes per subject to target scarring alopecia.
  Interventions: Device: Sciton HALO 1470nm Non-ablative laser

INTERVENTIONS:
Device: Sciton HALO 1470nm Non-ablative laser — Patients will be treated with the 1470nm non-ablative laser.

SUMMARY:
Single-center, open-label, baseline-controlled, pilot study evaluating the use of a Nonablative 1470 nm laser for the treatment of androgenetic alopecia and scarring alopecia.

DETAILED DESCRIPTION:
Single-center, open-label, baseline-controlled, pilot study evaluating the use of a Nonablative 1470 nm laser for the treatment of androgenetic alopecia and scarring alopecia. The study may enroll up to 10 participants looking for improvement in their hair loss. All participants will have biopsy-proven alopecia before enrollment. There will be two treatment arms with 5 participants in the androgenetic alopecia arm and 5 participants in the scarring alopecia arm. Multiple treatment areas of the scalp may be performed. Each subject will receive up to three treatments. Follow-up visits are planned for months 6, 9, 12, and 15. Standardized photography, hair density measurement of the treated scalp areas will be recorded Pre and Post Treatment at each visit. Measurement outcomes will be compared to baseline. During the initial visit, subjects who meet the study's eligibility criteria will receive the first treatment after signing informed consent form.

For this study, the investigators will use non-ablative HALO laser (1470nm) (Sciton). The non-ablative fractionated treatments with minimal downtime provide synergistic benefit of minimizing tissue damage while improving treatment tolerance and efficiency. The laser works by creating micro-channels in the dermis of the pilosebaceous unit, while leaving bridges of untouched tissue for improved permeability, faster healing, and enhanced delivery of topical treatments. The laser creates controlled zones of coagulation within the dermis. The parameters of the laser will be set according to optimal operation protocol and in accordance with guidelines set forth by Sciton. Each laser treatment will take approximately 10 to 15 minutes per subject. Pretreatment procedure will consist of topical anesthetic then cleaning of the affected area of the scalp with antiseptic, either 70% ethanol or 3% hydrogen peroxide. Post-treatment care will follow standard of care, including the application of topical betamethasone dipropionate cream 0.05% to the treated area. The U.S. Food and Drug Administration (FDA) has cleared the 1470 nm laser for dermatologic purposes. This study will use the laser off-label for the treatment of alopecia. This laser has been approved for the treatment of skin, however, it has not been tested for the treatment of androgenetic alopecia or scarring alopecia, thus this is a novel study to investigate its effectiveness

The follow up phase will consist of clinical assessments including before and after photographs graded by blinded observers and hair density evaluation using Canfield HairMetrix ® device. Subjects are instructed to inform clinical staff after the treatment if they experience any adverse events and will complete patient questionnaires, pain score, and self-assessment of hair growth.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, ≥ 18 years of age at time of informed consent, seeking treatment for hair loss
* Subject must voluntarily sign and date an IRB approved informed consent form
* Subjects with diagnosis of biopsy proven androgenetic alopecia or scarring alopecia with hair loss recorded over the past 6 months
* Subjects must have a stable hair loss treatment regimen with a plateau in results for at least 3 months
* Able to read, understand and voluntarily provide written informed consent
* Subject is determined to be healthy, non-smoker who agrees not to make any changes to their daily hair treatment regimen during the study
* Subjects able and willing to comply with the treatment protocol and follow-up schedule and requirements
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period

Exclusion Criteria:

* Subject does not have the capacity to consent to the study
* Subject has other types of alopecia of the scalp like alopecia areata
* Use of minoxidil or 5-alpha reductase inhibitors (i.e., finasteride, dutasteride) 3 months prior to screening date
* History of intralesional steroid injections to the scalp in the last 12 months
* Pregnant women
* Any medical condition that in the consideration of the investigator, would present an increased risk of a photosensitivity reaction to the subject
* Any previous surgical procedure in the treatment area in the past 12 months, or major surgery in the last 6 months
* Allergy or history of prior reaction to lidocaine
* History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection), and/or any history of systemic chemotherapy for prior 12 months
* History or current use of the following prescription medications:

  i. Immunosuppressive medications/biologics, 6 months prior to and during the study ii. Accutane or other systemic retinoids within the past twelve months
* Smoking or vaping in the past 12 months
* History of uncontrolled hyperlipidemia, diabetes mellitus, hepatitis, or bleeding disorders
* History of major depressive disorders or endocrine disorders including but not limited to; hypothyroidism, Hashimoto's thyroiditis, or hyperthyroidism

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Live and Photographic assessment of hair loss | month 1
  GAIS (Global Aesthetic Improvement Scale)- Scored from -3 greatly decreased in hair growth and density to 3 greatly increased in hair growth and density. A score of zero represents no change. This is the baseline assessment.
Hair density | month 1
  using Canfield HairMetrix imaging device; average number of hairs per follicular unit as baseline assessment
Hair counts | month 1
  using Canfield HairMetrix imaging device; hair count per cm squared as baseline assessment
Live and Photographic assessment of hair loss | Month 2
  GAIS (Global Aesthetic Improvement Scale)- Scored from -3 greatly decreased in hair growth and density to 3 greatly increased in hair growth and density. A score of zero represents no change.
Live and Photographic assessment of hair loss | Month 3
  GAIS (Global Aesthetic Improvement Scale)- Scored from -3 greatly decreased in hair growth and density to 3 greatly increased in hair growth and density. A score of zero represents no change.
Live and Photographic assessment of hair loss | Month 6
  GAIS (Global Aesthetic Improvement Scale)- Scored from -3 greatly decreased in hair growth and density to 3 greatly increased in hair growth and density. A score of zero represents no change.
Live and Photographic assessment of hair loss | Month 9
  GAIS (Global Aesthetic Improvement Scale)- Scored from -3 greatly decreased in hair growth and density to 3 greatly increased in hair growth and density. A score of zero represents no change.
Live and Photographic assessment of hair loss | Month 12
  GAIS (Global Aesthetic Improvement Scale)- Scored from -3 greatly decreased in hair growth and density to 3 greatly increased in hair growth and density. A score of zero represents no change.
Live and Photographic assessment of hair loss | Month 15
  GAIS (Global Aesthetic Improvement Scale)- Scored from -3 greatly decreased in hair growth and density to 3 greatly increased in hair growth and density. A score of zero represents no change.
Hair density | Month 6
  using Canfield HairMetrix imaging device; average number of hairs per follicular unit
Hair density | Month 9
  using Canfield HairMetrix imaging device; average number of hairs per follicular unit
Hair density | Month 12
  using Canfield HairMetrix imaging device; average number of hairs per follicular unit
Hair density | Month 15
  using Canfield HairMetrix imaging device; average number of hairs per follicular unit
Hair counts | month 6
  using Canfield HairMetrix imaging device; hair count per cm squared
Hair counts | month 9
  using Canfield HairMetrix imaging device; hair count per cm squared
Hair counts | month 12
  using Canfield HairMetrix imaging device; hair count per cm squared
Hair counts | month 15
  using Canfield HairMetrix imaging device; hair count per cm squared

SECONDARY OUTCOMES:
Subject Satisfaction | months 1
  1. Please choose the option that better represents the change in how your hair looks OVERALL in the area treated?
  2. Please choose the option that better represents the change in your hair THICKNESS in the area treated?
  3. Please choose the option that better represents the change in your hair SHEDDING/LOSS in the area treated?
  4. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
  5. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
     * -3 = Greatly decreased
     * -2 = Moderately decreased
     * -1 = Slightly decreased
     * 0 = No change
     * 1 = Slightly increased
     * 2 = Moderately increased
     * 3 = Greatly increased
Subject Satisfaction | month 2
  1. Please choose the option that better represents the change in how your hair looks OVERALL in the area treated?
  2. Please choose the option that better represents the change in your hair THICKNESS in the area treated?
  3. Please choose the option that better represents the change in your hair SHEDDING/LOSS in the area treated?
  4. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
  5. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
     * -3 = Greatly decreased
     * -2 = Moderately decreased
     * -1 = Slightly decreased
     * 0 = No change
     * 1 = Slightly increased
     * 2 = Moderately increased
     * 3 = Greatly increased
Subject Satisfaction | month 3
  1. Please choose the option that better represents the change in how your hair looks OVERALL in the area treated?
  2. Please choose the option that better represents the change in your hair THICKNESS in the area treated?
  3. Please choose the option that better represents the change in your hair SHEDDING/LOSS in the area treated?
  4. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
  5. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
     * -3 = Greatly decreased
     * -2 = Moderately decreased
     * -1 = Slightly decreased
     * 0 = No change
     * 1 = Slightly increased
     * 2 = Moderately increased
     * 3 = Greatly increased
Subject Satisfaction | month 6
  1. Please choose the option that better represents the change in how your hair looks OVERALL in the area treated?
  2. Please choose the option that better represents the change in your hair THICKNESS in the area treated?
  3. Please choose the option that better represents the change in your hair SHEDDING/LOSS in the area treated?
  4. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
  5. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
     * -3 = Greatly decreased
     * -2 = Moderately decreased
     * -1 = Slightly decreased
     * 0 = No change
     * 1 = Slightly increased
     * 2 = Moderately increased
     * 3 = Greatly increased
Subject Satisfaction | month 9
  1. Please choose the option that better represents the change in how your hair looks OVERALL in the area treated?
  2. Please choose the option that better represents the change in your hair THICKNESS in the area treated?
  3. Please choose the option that better represents the change in your hair SHEDDING/LOSS in the area treated?
  4. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
  5. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
     * -3 = Greatly decreased
     * -2 = Moderately decreased
     * -1 = Slightly decreased
     * 0 = No change
     * 1 = Slightly increased
     * 2 = Moderately increased
     * 3 = Greatly increased
Subject Satisfation | month 12
  1. Please choose the option that better represents the change in how your hair looks OVERALL in the area treated?
  2. Please choose the option that better represents the change in your hair THICKNESS in the area treated?
  3. Please choose the option that better represents the change in your hair SHEDDING/LOSS in the area treated?
  4. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
  5. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
     * -3 = Greatly decreased
     * -2 = Moderately decreased
     * -1 = Slightly decreased
     * 0 = No change
     * 1 = Slightly increased
     * 2 = Moderately increased
     * 3 = Greatly increased
Subject Satisfaction | month 15
  1. Please choose the option that better represents the change in how your hair looks OVERALL in the area treated?
  2. Please choose the option that better represents the change in your hair THICKNESS in the area treated?
  3. Please choose the option that better represents the change in your hair SHEDDING/LOSS in the area treated?
  4. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
  5. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
     * -3 = Greatly decreased
     * -2 = Moderately decreased
     * -1 = Slightly decreased
     * 0 = No change
     * 1 = Slightly increased
     * 2 = Moderately increased
     * 3 = Greatly increased

CONTACTS AND LOCATIONS:
Overall Officials: Kseniya Kobets, MD, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Montefiore Einstein Advanced Care, Elmsford, New York, United States

IPD SHARING:
Plan to Share IPD: No